CLINICAL TRIAL: NCT02785172
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study to Compare the Safety and Efficacy of IDP-118 Lotion to Ultravate® in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy of IDP-118 Lotion to Ultravate® in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-118A-203
Record Dates: First submitted 2016-04-26; First posted 2016-05-27 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — halobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IDP-118 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-118 Lotion
- Ultravate Cream (Active Comparator): Cream
  Interventions: Drug: Ultravate Cream
- IDP-118 Vehicle Lotion (Active Comparator): Lotion
  Interventions: Drug: IDP-118 Vehicle Lotion
- IDP-118 Vehicle Cream (Active Comparator): Cream
  Interventions: Drug: IDP-118 Vehicle Cream

INTERVENTIONS:
Drug: IDP-118 Vehicle Lotion — Vehicle
  Other Names: Lotion
  Arms: IDP-118 Vehicle Lotion
Drug: IDP-118 Vehicle Cream — Vehicle
  Other Names: Cream
  Arms: IDP-118 Vehicle Cream
Drug: IDP-118 Lotion — Lotion
  Other Names: Lotion
  Arms: IDP-118 Lotion
Drug: Ultravate Cream — Cream
  Other Names: Ultravate
  Arms: Ultravate Cream

SUMMARY:
Safety and Efficacy of IDP-118 Lotion to Ultravate® Cream, in the Treatment of Plaque Psoriasis

DETAILED DESCRIPTION:
A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study to Compare the Safety and Efficacy of IDP-118 Lotion to Ultravate® Cream, in the Treatment of Plaque Psoriasis

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Has an area of plaque psoriasis appropriate for topical treatment that covers a BSA (Body Surface Area) of at least 3%, but no more than 12%. The face, scalp, palms, soles, axillae, and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an IGA (Investigators Global Assessment) score of 3 or 4. (The face, scalp, palms, soles, axillae, and intertriginous areas are to be excluded in this assessment, if psoriasis is present.)
* If female and of childbearing potential, must have a negative urine and serum pregnancy test at the Screening visit and negative urine pregnancy at Baseline visit prior to randomization.
* Subject is willing to comply with study instructions and return to the clinic for required visits.

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half-lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, MD, Study Director — Valeant Pharmaceuticals; Binu Alexander, Study Director — Valeant Pharmaceuticals
Locations (14):
- United States (14):
  - Valeant Site 12, Fullerton, California
  - Valeant Site 04, La Mesa, California
  - Valeant Site 03, San Diego, California
  - Valeant Site 09, San Diego, California
  - Valeant Site 05, Lauderdale Lakes, Florida
  - Valeant Site 02, Miami, Florida
  - Valeant Site 07, Fridley, Minnesota
  - Valeant Site 08, Chapel Hill, North Carolina
  - Valeant Site 06, Columbus, Ohio
  - Valeant Site 13, Mt. Pleasant, South Carolina
  - Valeant Site 11, Katy, Texas
  - Valeant Site 10, San Antonio, Texas
  - Valeant Site 01, Sugar Land, Texas
  - Valeant Site 14, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IDP-118 Lotion | Ultravate Cream | IDP-118 Vehicle Lotion | IDP-118 Vehicle Cream
Started | 61 | 63 | 16 | 14
Completed | 61 | 62 | 15 | 14
Not Completed | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDP-118 Lotion | Ultravate Cream | IDP-118 Vehicle Lotion | IDP-118 Vehicle Cream | Total
Number analyzed (Participants) | 61 | 63 | 16 | 14 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (13.81) | 49.5 (13.47) | 48.3 (11.63) | 52.5 (9.37) | 50.36 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 6 | 6 | 62
  Male | 32 | 42 | 10 | 8 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Treatment Success
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the Investigator's Global Assessment (IGA) score and an IGA score equating to "clear" or "almost clear". The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion | Ultravate Cream | IDP-118 Vehicle Lotion | IDP-118 Vehicle Cream
Number analyzed (Participants) | 61 | 63 | 16 | 14
percentage of participants | 32.79 | 33.97 | 0 | 7.14

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were collected from participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-Baseline safety assessment (Safety Population).
Arm/Group | IDP-118 Lotion | Ultravate Cream | IDP-118 Vehicle Lotion | IDP-118 Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/62 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/61 | 0/62 | 0/15 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=61) | Ultravate Cream (N=62) | IDP-118 Vehicle Lotion (N=15) | IDP-118 Vehicle Cream (N=14)
Application site atrophy (General disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.h